CLINICAL TRIAL: NCT07032792
Title: Factor VIII Inhibitor Bypass Activity (FEIBA) Versus Fresh Frozen Plasma As First Line Therapy For Bleeding After Cardiac Surgery
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0293
Record Dates: First submitted 2025-04-21; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Disease; Surgery; Bleeding
MeSH Terms: conditions — Heart Diseases; Hemorrhage | interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FEIBA (Experimental)
  Interventions: Drug: FEIBA
- FFP (Active Comparator)
  Interventions: Drug: FFP

INTERVENTIONS:
Drug: FEIBA — Subjects randomized to FEIBA will receive up to 2 vials of 500U of FEIBA through a preexisting central line at a rate that does not exceed 2 units per kg of body weight per minute for the study intervention.
  Arms: FEIBA
Drug: FFP — Subjects randomized to FFP will receive up to 2 units of FFP intravenously through a preexisting central line.
  Arms: FFP

SUMMARY:
Coagulopathic-induced bleeding after cardiopulmonary bypass in cardiac surgery patients is common and is associated with adverse outcomes in cardiac surgery. The hypothesis of the study is that FEIBA will be a more effective treatment than standard of care (FFP) in cardiac surgery patients who have coagulopathic-induced bleeding. This study is being conducted to determine the efficacy of FEIBA versus FFP as first line therapy in correcting coagulopathic induced microvascular bleeding in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 years or above
* Undergoing nonemergent non-coronary cardiac surgery with the use of cardiopulmonary bypass
* Patient with microvascular bleeding requiring factor transfusion as deemed by the patient care team

Exclusion Criteria:

* Contraindication to the administration of FEIBA or known anaphylactic or severe hypersensitivity reaction to FEIBA or any of its components
* Disseminated intravascular coagulation
* Acute thrombosis or embolism, including myocardial infarction
* Pregnancy
* Patients that are not able or do not want to consent for themselves
* Patients with known coagulation disorders
* Patients who received coronary artery bypass surgery
* Patients who received transplants or ventricular assist devices
* Patients on extracorporeal membrane oxygenator support
* Patients with heparin induced thrombocytopenia
* Patients who do not wish to receive blood products even when it is deemed medically necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Total post-treatment pRBC transfusion within 24 hours of surgery | 24 hours

SECONDARY OUTCOMES:
Total pRBC transfusion after administration of study drug | From time of administration of study drug until time of discharge or up to 3 months, whichever comes first.
Total units of posttreatment platelet transfusion within 24 hours of surgery | 24 hours
Total units of posttreatment cryoprecipitate transfusion within 24 hours of surgery | 24 hours
Total units of FEIBA given within 24 hours of surgery | 24 hours
Total units of Fresh Frozen Plasma (FFP) given within 24 hours of surgery | 24 hours
Total mLs of chest tube output within 12 hours of surgery | 12 hours
  This is being assessed as chest tube output may be an indicator of ongoing bleeding
Incidence of adverse postoperative events | Perioperative
  This can include thrombotic events, acute kidney injury, reoperation for bleeding, prolonged intubation, atrial fibrillation, anaphylaxis.
Length of intubation | Perioperative
Length of hospital stay | From date of hospital admission until date of discharge or up to 3 months, whichever comes first.
30-day mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pey-Jen Yu, Principal Investigator — Northwell Health
Locations (1):
- North Shore University Hospital, Manhasset, New York, United States